

### ANNEX 1

#### INFORMED CONSENT

First of all, I would like to **thank you for your collaboration** in this study on transcutaneous stimulation. Without your help this study could not be carried out. Thank you for your collaboration.

## 1. What is this study and what does it aim to achieve?

This study aims to quantify sleep quality, symptom perception and quality of life in subjects with urinary incontinence. The study will be divided into two randomised groups, one group will receive the NXSignal application and the other group will receive electrostimulation of the posterior tibial nerve.

There are currently various types of treatment for overactive bladder, however, physiotherapy treatment using neuromodulation techniques has been found to offer good results for patients with overactive bladder. Participation in the study is voluntary, no one is obliged to participate. At the same time, anyone can leave the study at any time without having to give any explanation.

#### Benefits and risks.

The study does not pose any potential risk to the participants. As a post-treatment effect, in some cases of particularly sensitive persons, reddening of the skin in the area of the electrodes may occur after the treatment; the redness usually disappears within a few minutes after the treatment. This study is approved by the Valencia University ethical committee (Cod. 2025-FIS-3870878).

# 3. Confidentiality of data

In accordance with Spanish Law 15/1999 on the Protection of Personal Data, the personal data required (sex, age, etc.) are those necessary to carry out the study correctly. None of this data will be disclosed to external persons. Your participation is anonymous. However, your names will be recorded on a checklist that will be kept by the principal investigator and will only be used when necessary. In accordance with current law, you have the right of access to your personal data and, if duly justified, the right to rectify and delete them. If you so wish, you should request this from the researcher in charge of your care. The results of the study may be communicated to the health authorities and, eventually, to the scientific community through congresses and/or publications.

| I, (patient's name) | |
|---|---|
| I have read the information sheet given to me, I have been able to ask the necessary questions about the study and I have voluntarily agreed to participate in this study. | |
| Date | Participant's signature (handwritten by participant) |
| The principal investigator of these study | y: Paloma Blasco-Sonora. (approved date 04.04.2025) |